CLINICAL TRIAL: NCT00241982
Title: Long-Circulating Liposomal Prednisolone Versus Pulse Intramuscular Methylprednisolone in Patients With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Utrecht University (Other)
Responsible Party: Dr. Pilar Barrera, Radboud University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: liposomal prednisolone
Record Dates: First submitted 2005-10-18; First posted 2005-10-19 (Estimated); Last update posted 2008-05-30 (Estimated); Status verified 2008-05

CONDITIONS: Rheumatoid Arthritis
Keywords: rheumatoid arthritis; long circulating liposomes
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: long-circulating liposomal prednisolone

SUMMARY:
Trial to study the safety of a single, intravenous administration of long-circulating liposomal prednisolone disodium phosphate in patients with active rheumatoid arthritis.

DETAILED DESCRIPTION:
A proof of concept, dose-escalating trial to study the safety of a single, intravenous administration of long-circulating liposomal prednisolone disodium phosphate in patients with active rheumatoid arthritis.

Secondary goals: To compare the therapeutic effect of this intervention with that of a single intramuscular administration of 120 mg methylprednisolone (Depo-Medrol, Pharmacia). The latter is commonly used in the clinics as bridging therapy. To assess the effect of these interventions at the synovial tissue level.

On the longer term, the goal of liposomal corticosteroids is to achieve an increased efficacy/safety ratio compared to standard treatment with free corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

In order to be enrolled in the study a patient must:

Be aged 18 years or older Fulfill the revised 1987 ARA criteria for the classification of RA Have an active RA as defined by a Modified Disease Activity Score (DAS28) of more than 3.2 Have been on stable treatment with disease modifying anti-rheumatic drugs within 12 weeks prior to trial initiation Be able and willing to give voluntary written informed consent The indication for bridging therapy with systemic corticosteroids has been established by the caring rheumatologist -

Exclusion Criteria:

The patient must not Have been treated with oral corticosteroids within 2 weeks prior to baseline or with intraarticular or intramuscular corticosteroids within 8 weeks prior to baseline Have diabetes mellitus or abnormal renal, liver or haematological tests Have a clinically severe or unstable medical condition involving cardiac, pulmonary, liver and endocrine disorders or malignancies Have a previous history of bleeding or infectious disorders Be currently pregnant or breastfeeding

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2005-10; Primary Completion 2008-03 (Actual); Study Completion 2008-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: P. Barrera, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud University Nijmegen Medical Centre, Nijmegen, Gelderland, Netherlands